CLINICAL TRIAL: NCT00620620
Title: Safety, Tolerability, and Pharmacokinetics of a Single Dose of Staccato® Zaleplon for Inhalation in Healthy Volunteers
Brief Title: Staccato Zaleplon Single Dose Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMDC-007-101; 17 December 2007
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2013-07

CONDITIONS: Healthy
Keywords: Healthy adult volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Inhaled Placebo (Placebo Comparator): Staccato Placebo
  Interventions: Drug: Inhaled placebo
- Inhaled Zaleplon 0.5 mg (Experimental): Staccato Zaleplon 0.5 mg
  Interventions: Drug: Inhaled Zaleplon 0.5 mg
- Inhaled Zaleplon 1 mg (Experimental): Staccato Zaleplon 1 mg
  Interventions: Drug: Inhaled Zaleplon 1 mg
- Inhaled Zaleplon 2 mg (Experimental): Staccato Zaleplon 2 mg
  Interventions: Drug: Inhaled Zaleplon 2 mg
- Inhaled Zaleplon 4 mg (Experimental): Staccato Zaleplon 4 mg
  Interventions: Drug: Inhaled Zaleplon 4 mg

INTERVENTIONS:
Drug: Inhaled placebo — Inhaled Staccato Placebo
  Other Names: Staccato Placebo
  Arms: Inhaled Placebo
Drug: Inhaled Zaleplon 0.5 mg — Inhaled Staccato Zaleplon 0.5 mg
  Other Names: Staccato Zaleplon 0.5 mg
  Arms: Inhaled Zaleplon 0.5 mg
Drug: Inhaled Zaleplon 1 mg — Inhaled Staccato Zaleplon 1 mg
  Other Names: Staccato Zaleplon 1 mg
  Arms: Inhaled Zaleplon 1 mg
Drug: Inhaled Zaleplon 2 mg — Inhaled Staccato Zaleplon 2 mg
  Other Names: Staccato Zaleplon 2 mg
  Arms: Inhaled Zaleplon 2 mg
Drug: Inhaled Zaleplon 4 mg — Inhaled Staccato Zaleplon 4 mg
  Other Names: Staccato Zaleplon 4 mg
  Arms: Inhaled Zaleplon 4 mg

SUMMARY:
The purpose of the study is to determine the safety, tolerability and pharmacokinetics of zaleplon delivered by the Staccato thermal aerosol system in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 to 55 years, inclusive who are in good general health

Exclusion Criteria:

* Subjects with a history of allergy or intolerance to zaleplon. Subjects who have any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Examine the tolerability and safety of Staccato Zaleplon in a healthy volunteer population; | Single dose

SECONDARY OUTCOMES:
Establish the plasma level-time profile (pharmacokinetics) of zaleplon in the target therapeutic range following single Staccato Zaleplon doses | single dose

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Spyker, MD, Study Director — Alexza Pharmaceuticals, Inc.
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com

REFERENCES:
- [Background] Avram MJ, Spyker DA, Kehne JH, Cassella JV. The pharmacokinetics and pharmacodynamics of zaleplon delivered as a thermally generated aerosol in a single breath to volunteers. J Clin Pharmacol. 2013 Feb;53(2):140-50. doi: 10.1177/0091270012436886. PMID 23436259